CLINICAL TRIAL: NCT02143232
Title: Postop Home Monitoring After Joint Replacements (POHM)
Brief Title: Post Op Home Monitoring After Joint Replacements
Acronym: POHM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: The Ottawa Hospital Academic Medical Association (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20130412-01H
Record Dates: First submitted 2014-05-12; First posted 2014-05-21 (Estimated); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Total Knee Replacement; Total Hip Replacement
Keywords: knee replacement; hip replacement; patient monitor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Remote patient monitoring (Telus RPM) (Experimental): The remote monitoring device (Telus RPM) is used by every patient in the study post operatively at home.
  Interventions: Device: remote patient monitoring (Telus RPM)

INTERVENTIONS:
Device: remote patient monitoring (Telus RPM) — All joint replacement patients in the study will use the same type of remote patient monitor for 4 days post operation at home.
  Other Names: Telus RPM

SUMMARY:
The investigators propose to deploy an interactive device to monitor the patient's recovery and vital signs at home after joint replacements. These will be early discharge patients on the same day or the next morning. The goal will be to support early discharges by creating a safe, controlled, and monitored environment at home.

DETAILED DESCRIPTION:
1. Background and rationale. According to the latest Canadian Census, seniors aged 65 or over have increased in number by 609,810 from 13.7% of the population in 2006 to 4,945,060, or 14.8% in 2011. In Ontario, in 2001, there were 8,000 total hip replacements (THR) and 11,000 total knee replacements (TKR); in 2016, the projection is 20,000 THR and 54,000 TKR, assuming age-specific rates remain the same(1). At The Ottawa Hospital (TOH), we have already witnessed the pressure on bed management due to the increasing case volume. As a solution, we have successfully organized early discharges (EDc), on the same day, in select patients after unicompartment arthroplasty in order to reduce the length of stay (LOS)(2). Since then, we have discharged select major joint replacement patients on the same day or after overnight stay on multimodal analgesia.

   A remote patient monitoring interactive system for chronic disease care. This monitor allows telephone or wireless connectivity with the patient and is equipped with NIBP (non-invasive blood pressure), HR (heart rate), and SpO2 (pulse oximetry) measurements that the patient or a caretaker could use at home. It generates regular reminders for the patient to measure his/her NIBP, HR, glucose levels if appropriate and SpO2 as well as answer a scripted questionnaire for pain. Results and alerts are then transmitted to the healthcare team. The system has never been deployed in an acute care or post-op environment. We propose therefore to conduct a feasibility study on early discharge patients after unicompartment or total joint replacements, deploying the Telus interactive RPM with our existing early discharge care path.
2. Methods This is a feasibility study to allow planning for a larger future study to prove the above hypothesis.

A sample size of 54 is sufficient to yield a one-sided 95% confidence interval estimate around our primary outcome measure (proportion of successful transmissions) with a lower bound exceeding the cutpoint for feasibility of 90%, assuming a proportion of 95% successful transmission. Recruitment will be at the orthopedic clinics, using the approved OHRI "Consent for Personal Health Information Review for Research Purposes" obtained through a member of the circle of care. Informed consent will be obtained at the General Pre-Admission Unit (PAU) by the research assistant after eligibility has been determined. A screening process for unicompartment knee arthroplasty and care path for same day discharge is currently in place. For this study, care paths for same day / early discharge for total hip and knee arthroplasty will be confirmed. Theses care paths will include home visits by nursing and physio through the Community Care Access Centre (CCAC).

Patients who satisfy the early discharge criteria will be approached. After informed consent the use of the remote patient monitoring device will be demonstrated . prior to discharge, after ensuring that the patient has achieved the defined outcomes of the care path, the functionalities of the device will be reviewed with the patient and care-taker. The patient will be given the monitor to bring home and set up. If required a member of the study team will assist you with the set up and use of the device This may require a home visit. CCAC visit will be as outlined in the care path and at the latest by the next day. Monitoring will be continued for 4 days at home.The system will be repatriated to TOH for cleaning and preventative maintenance.

Post-operative complications will be documented at Day 4 and with a followup phone call at 30 days, including POMI (postoperative myocardial infarction),CHF (congestive heart failure),DVT (deep vein thrombosis), PE (pulmonary embolism)pneumonia, cardiac dysrhythmia requiring treatment, wound dehiscence, and surgical site infections (SSI). The patient satisfaction questionnaire will include concerns with the RPM as well as the healthcare team response and will be completed by the patient using the patient monitoring system within 48 hours after the monitoring is completed.A followup phone call will occur at Day 30. Results from this feasibility study will be used to plan a future large-scale randomized controlled trial to evaluate effectiveness and safety of the above.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective hip or knee arthroplasty
* Expected LOS ≤ 1 day
* Age 50 - 80 years
* Revised Cardiac Risk Index (RCRI) ≤ Class 2
* Available and able care-takers at home to assist the patient upon discharge during the early postoperative recovery phase.

Exclusion Criteria:

* ASA IV (American Association of Anesthesiology) classification
* COPD (chronic obstructive pulmonary disease) with FEV1 ≤ 1; (forced expiratory volume) OSA (obstructive sleep apnea)
* Patient or family reluctance to participate in early discharge
* Undiagnosed or on-going medical condition at time of discharge
* Previous participation in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2014-04; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Successful transmission of ≥ 90% of patients' assessments from the patient station to the clinical station using the remote monitoring system. | Home Monitoring followup after hospital discharge for 4 days, 4 times during the day and as needed.
  The patient will do a measure of his/her blood pressure, heart rate,oxygen saturation, glucose levels (if appropriate) and pain assessment and this will be transmitted to a clinical station for observation by a clinical /medical person. Such a system is interactive, providing support to the patient at home, with reminders for medications, glucose control,blood pressure control, and a conduit to report problems such as pain and those associated with the surgical incision. Patients upon early discharge may also feel isolated, especially if there are questions on surgical and medical management issues or pain control. The alert system provides a safe and reliable communications channel for the patient.
  .

SECONDARY OUTCOMES:
Difference in the incidence of unplanned readmissions or unplanned visits to the ED compared to 54 patients from a historical cohort 2010 - 2011 matched in age, sex, and procedures | The cohort selected will be from 2010 to 2011. (up to 1 year)
  Chart Review

CONTACTS AND LOCATIONS:
Overall Officials: Homer Yang, MD, Principal Investigator — Clinical Investigator
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dervin GF, Madden SM, Crawford-Newton BA, Lane AT, Evans HC. Outpatient unicompartment knee arthroplasty with indwelling femoral nerve catheter. J Arthroplasty. 2012 Jun;27(6):1159-65.e1. doi: 10.1016/j.arth.2012.01.009. Epub 2012 Mar 28. PMID 22459126
- [Derived] Yang H, Dervin G, Madden S, Fayad A, Beaule P, Gagne S, Crossan ML, Wheeler K, Afagh M, Zhang T, Taljaard M. Postoperative Home Monitoring After Joint Replacement: Retrospective Outcome Study Comparing Cases With Matched Historical Controls. JMIR Perioper Med. 2018 Nov 5;1(2):e10169. doi: 10.2196/10169. PMID 33401365
- [Derived] Yang H, Dervin G, Madden S, Beaule PE, Gagne S, Crossan ML, Fayad A, Wheeler K, Afagh M, Zhang T, Taljaard M. Postoperative Home Monitoring After Joint Replacement: Feasibility Study. JMIR Perioper Med. 2018 Sep 5;1(2):e10168. doi: 10.2196/10168. PMID 33401364